CLINICAL TRIAL: NCT04967820
Title: Burn-out Among Chinese Anaesthesiologist After COVID-19 Pandemic Peak and Its Protective Factor: a National Survey
Brief Title: Burn-out Among Chinese Anaesthesiologist After COVID-19 Pandemic Peak and Its Protective Factor： a National Survey
Status: Completed | Type: Observational
Sponsor: Huang YuGuang (Other)
Collaborators: Chinese Society of Anesthesiology (Unknown)
Responsible Party: Sponsor-Investigator, Huang YuGuang, head of anaesthesiology department, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: CSAnationalsurveyburnout
Record Dates: First submitted 2021-07-02; First posted 2021-07-20 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: resilience and institutional support — psychological inherent resilience and institutional support during COVID-19 outbreak

SUMMARY:
The investigators proposed a national representative survey to collect data of socio-demographic characteristics, level of exposure to COVID-19, depression，anxiety， ptsd， burnout and resilience of working anaesthesiologists across mainland China for the following purpose

1. Explore the current burn-out rate of Chinese anaesthesiologists and compared it with data acquired in 2015；
2. Explore the perceived covid-19 exposure of COVID-19 among Chinese anaesthesiologist.
3. Explore rate of burnout, anxiety, depression, PTSD symptoms experienced by the participants
4. Explore the protective psychosocial characteristics of burnout. (resilience)
5. See whether covid-19 exposure contribute to higher burn out rate.

ELIGIBILITY:
Inclusion Criteria:

working anaesthesiologist in mainland China

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: working anaesthesiologist in mainland China
Sampling Method: Non-Probability Sample
Enrollment: 6631 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Burnout | data will be retrieved and recored 1 week after survey distribution
  Burnout level will be measured by Maslach Burnout Inventory-Human Service Survey

OTHER OUTCOMES:
Post-Traumatic Stress Disorder | data will be retrieved and recored 1 week after survey distribution
  The Impact of Events Scale-Revised (IES-R) is a self-reporting tool widely used in the field of psychological impact and has been proven to be suitable for the Chinese population
Resilience | data will be retrieved and recored 1 week after survey distribution
  10-item Connor-Davidson Resilience Scale (CD-RISC-10) was used to assess resilience.
Depressive symptoms | data will be retrieved and recored 1 week after survey distribution
  The Patient Health Questionnaire-9 (PHQ-9) was included to assess depressive symptoms.
Anxiety | data will be retrieved and recored 1 week after survey distribution
  Anxiety level will be evaluated by GAD-7 Anxiety Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Che L, Ma S, Zhang YL, Huang Y. Burnout Among Chinese Anesthesiologists After the COVID-19 Pandemic Peak: A National Survey. Anesth Analg. 2023 Aug 1;137(2):392-398. doi: 10.1213/ANE.0000000000006298. Epub 2022 Dec 2. PMID 36729947